CLINICAL TRIAL: NCT01383395
Title: Effect of Cilostazol on the Pharmacokinetics of Simvastatin in Healthy Adult Subjects
Brief Title: Effect of Cilostazol on the Pharmacokinetics of Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Inje University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-04-070
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — Simvastatin; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- simvastatin/cilostazol (Experimental): simvastatin 40 mg on day 1 and 6, cilostazol 100 mg from day 2 to day 6
  Interventions: Drug: simvastatin/cilostazol

INTERVENTIONS:
Drug: simvastatin/cilostazol

SUMMARY:
To evaluate the effect of cilostazol on the pharmacokinetics of simvastatin in healthy adult subjects.

DETAILED DESCRIPTION:
Eligibility for participation of this study was determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study were admitted to the Clinical Trials Center, Samsung Medical Center on the day before dosing, and they were overnight-fasted from 10 p.m. of Day -1. Subjects were dosed simvastatin 40 mg orally around at 9 a.m. of Day 1. Subjects performed scheduled procedures including clinical laboratory tests and pharmacokinetic samplings for simvastatin. Subjects were dosed cilostazol 100 mg in the morning on Day 2 and discharged, and visited Clinical Trials Center on Day 3, Day 4 and Day 5 for the oral administration of cilostazol 100 mg. Subjects was admitted in the evening on day 5 and dosed simvastatin 40 mg plus cilostazol 100 mg concomitantly and scheduled pharmacokinetic sampling for simvastatin was performed. Next morning (Day 7), subjects were discharged

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 48 years
* A body mass index (BMI) in the range 19-27 kg/m2
* Provide written informed consent after being fully informed about the study procedures
* Subject without any congenital or chronic disease and with no pathologic symptom in the physical examination
* Determined eligible in the ECG, clinical laboratory tests and urinalysis

Exclusion Criteria:

* Use of medication which induces or inhibits drug metabolizing enzyme (CYP3A4 etc.) within 30 days prior to drug dosing
* Use of medication within 10 days before first dose
* Abnormal diet that can influence on tlhe ADME of drugs (grapefruit juice etc.)
* Presence or history of clinically significant allergic disease, alcohol abuse, drug hypersensitivity
* Whole blood donation during 60 days before the study
* Participation in other clinical trial within 90 days prior to scheduled study drug administration
* Subject judged not eligible for study participation by investigator

Ages: 20 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of simvastatin | 7 days
  Plasma concentration of simvastin on day 1 and day 6

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center Clinical Trial Center, Seoul, South Korea